CLINICAL TRIAL: NCT02201667
Title: An Open-label Study Evaluating the Acute Efficacy of Treatment With Ticagrelor Versus Clopidogrel on Myocardial Tissue-level Perfusion Assessed by TMPFC and MRI in Patients With High-risk NSTE-ACS Undergoing Early PCI（EARLY-MYO II）
Brief Title: Efficacy of Ticagrelor vs Clopidogrel in High-risk NSTE-ACS Patients Undergoing Early PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0208
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Acute Coronary Syndrome
Keywords: non-ST elevation acute coronary syndrome; myocardial perfusion; magnetic Resonance Imaging; antiplatelet
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor group (Experimental): Patients wil be given 180 mg loading dose of ticagrelor and 300mg loading dose of aspirin followed by PCI, then will receive 90 mg ticagrelor twice daily with aspirin maintenance dose to 30 days after randomization.
  Interventions: Drug: Ticagrelor; Drug: Aspirin; Procedure: PCI
- Clopidogrel group (Active Comparator): Patients will be given clopidogrel 300mg loading dose and 300mg loading dose of aspirin followed by PCI, then will receive 75mg clopidogrel once with aspirin maintenance dose to 30 days after randomization.
  Interventions: Drug: clopidogrel; Drug: Aspirin; Procedure: PCI

INTERVENTIONS:
Drug: Ticagrelor — 180-mg loading dose followed by 90mg twice daily for 30 days
  Other Names: BRILINTA
  Arms: Ticagrelor group
Drug: clopidogrel — 300-mg loading dose followed by 75mg once daily for 30 days.
  Other Names: Plavix
  Arms: Clopidogrel group
Drug: Aspirin — 300mg loading dose aspirin and followed by 100mg once daily
  Other Names: Aspirin Enteric Coated Tablets
Procedure: PCI — PCI is performed according to indication for early PCI according to 2012 Chinese NSTE-ACS guideline recommendation

SUMMARY:
The goal of acute coronary syndrome (ACS) therapy is to successfully restore both epicardial blood flow and myocardial perfusion. Percutaneous coronary intervention (PCI) has been documented as being the most effective method for restoration of epicardial blood flow. However, epicardial blood flow does not necessarily equate to myocardial perfusion. Clopidogrel binds irreversibly to platelet P 2 Y 12 receptors to inhibit platelet aggregation, with main limitations of slow onset, prevention of recovery of platelet functions, and interindividual variability. Clinical pharmacology and early dose-finding studies suggested a faster onset and greater and more consistent inhibition of platelet aggregation (IPA) with ticagrelor compared with clopidogrel. Two currently main methods of angiographic assessment of myocardial perfusion includes thrombolysis in myocardial infarction(TIMI) myocardial perfusion grading (TMPG) and myocardial blush grading (MBG). These established myocardial perfusion parameters have been widely used in various important trials and are reported to be highly useful in predicting clinical outcomes. However, visual assessment of these methods is categorical, subjective, and operator dependent of contrast in the myocardium using cine-angiographic frame-counting, was developed by the investigators' center to quantify myocardial tissue- level perfusion and was proved to be a predictive value on clinical prognosis.

Thus, the investigators aim to initiate an open-label study evaluating the acute efficacy of treatment with ticagrelor versus clopidogrel on myocardial tissue-level perfusion assessed by Myocardial Perfusion Frame Count(TMPFC) and magnetic resonance imaging (MRI) in patients with high-risk non-ST elevation acute coronary syndrome (NSTE-ACS) undergoing early percutaneous coronary intervention (PCI) .

The investigators hypothesize that compared with clopidogrel, ticagrelor can significantly improve myocardial perfusion assessed by Myocardial Perfusion Frame Count(TMPFC) in high-risk non-ST elevation acute coronary syndrome (NSTE-ACS) patients undergoing early percutaneous coronary intervention (PCI), without additional increased major bleeding.

DETAILED DESCRIPTION:
The goal of acute coronary syndrome (ACS) therapy is to successfully restore both epicardial blood flow and myocardial perfusion. Percutaneous coronary intervention (PCI) has been documented as being the most effective method for restoration of epicardial blood flow. However, epicardial blood flow does not necessarily equate to myocardial perfusion; not every patient with thrombolysis in myocardial infarction(TIMI) 3 flow after successful percutaneous coronary intervention (PCI) achieves effective myocardial tissue-level perfusion. Although epicardial thrombolysis in myocardial infarction(TIMI) 3 flow could be restored in >90% of acute coronary syndrome (ACS) patients undergoing percutaneous coronary intervention (PCI) , normalization of myocardial perfusion was achieved less frequently, with detrimental impacts on survival.

Clopidogrel, the most widely used antiplatelet agent in acute coronary syndrome (ACS), is a thienopyridine prodrug, which is inactive until in undergoes biotransformation into its active metabolite, which then binds irreversibly to platelet P 2 Y 12 receptors. This irreversible binding means that the receptors are inhibited for the lifespan of the platelet. The main limitations of clopidogrel administration include slow onset, prevention of recovery of platelet functions, and interindividual variability.

Clinical pharmacology and early dose-finding studies suggested a faster onset and greater and more consistent inhibition of platelet aggregation (IPA) with ticagrelor compared with clopidogrel. ONSET/OFFSET study showed that in patients with stable coronary artery disease on aspirin, ticagrelor demonstrates a rapid onset of pharmacological effect, as demonstrated by a mean platelet aggregation (IPA) for ticagrelor at 0.5 h after 180 mg loading dose of about 41%, with the maximum platelet aggregation (IPA) effect of 87.9-89.6% by 2-4 hours post dose. A total of 90% of patients had final extent Inhibition of platelet aggregation (IPA) >70% by 2 h post-dose. The high inhibition of platelet aggregation (IPA) effect of ticagrelor (between 87% and 89%) was maintained for 2-8 hours. Ticagrelor might overcome the slow-onset limitation of clopidogrel and bring extra benefit for improving myocardial perfusion in the acute phase of acute coronary syndrome (ACS) when undergoing early percutaneous coronary intervention (PCI).

Currently, there are two main methods of angiographic assessment of myocardial perfusion: Thrombolysis in myocardial infarction (TIMI) myocardial perfusion grading (TMPG), described by Gibson et al. and myocardial blush grading (MBG), described by Van't Hof et al. These established myocardial perfusion parameters, myocardial perfusion grading (TMPG), and myocardial blush grading (MBG), have been widely used in various important trials and are reported to be highly useful in predicting clinical outcomes. However, visual assessment of these methods is categorical, subjective, and operator dependent. Thrombolysis in myocardial infarction(TIMI) Myocardial Perfusion Frame Count (TMPFC), a novel and objective method that measures the filling and clearance of contrast in the myocardium using cine-angiographic frame-counting, was developed by the investigators' center to quantify myocardial tissue- level perfusion and was proved to be a predictive value on clinical prognosis.

Thus, the investigators aim to initiate an open-label study evaluating the acute efficacy of treatment with ticagrelor versus clopidogrel on myocardial tissue-level perfusion assessed by Myocardial Perfusion Frame Count (TMPFC) and magnetic resonance imaging (MRI) in patients with high-risk non-ST elevation acute coronary syndrome (NSTE-ACS) undergoing early percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Men or women > 18 years of age, with documented evidence of non-ST segment elevation Acute Coronary Syndrome(ACS) in the 24 hours before randomisation;
3. Hospitalized for high-risk non-ST segment elevation Acute Coronary Syndrome(ACS)(GRACE risk score>140) with indication for early percutaneous coronary intervention (PCI) according to 2012 Chinese non-S T segment elevation Acute Coronary Syndrome(ACS) guideline recommendation.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Evidence of cardiac rupture;
2. History of major hemorrhage (intracranial, gastrointestinal, etc.);
3. Active pathological bleeding;
4. Acute or chronic hematologic disorder including a Hemoglobin less than 10 g/L or a platelet count less than 10×109/L before procedure;
5. Contraindication against the use of clopidogrel and ticagrelor;
6. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
7. Severe complication 7.1 Other diseases with life expectancy ≤12 months; 7.2 Any history of Severe renal or hepatic dysfunction(hepatic failure, cirrhosis, portal hypertension and active hepatitis); Neutropenia, thrombocytopenia ; Known acute pancreatitis; 7.3 Arterial aneurysm, arterial/venous malformation and aorta dissection;
8. Complex heart condition 8.1 PCI within previous 1 month or Previous coronary-artery bypass surgery(CABG); 8.2 History of myocardial infarction; 8.3 Previously known multivessel coronary artery disease not suitable for percutaneous coronary intervention (PCI);
9. Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 30 days;
10. Treatment with anticoagulants;
11. Pregnancy or lactating;
12. Body weight <40kg or >125kg;
13. Known hypersensitivity to any drug that may appear in the study;
14. Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
TIMI Myocardial Perfusion Frame Count (TMPFC) | Within 0 to 24 hours after randomization
  The Myocardial Perfusion Frame Count (TMPFC) is developed to standardize and quantify myocardial perfusion by timing the filling and clearance of contrast in the myocardium using cine-angiographic frame-counting. The first frame of Myocardial Perfusion Frame Count (TMPFC) is defined as the frame that clearly demonstrates the first appearance of myocardial blush beyond the infarct-related artery (IRA) (F1). The last frame of Myocardial Perfusion Frame Count (TMPFC) is then defined as the frame where contrast or myocardial blush disappears (F2). TMPFC is therefore F2-F1 frame counts at filming rate of 15frames/sec.

SECONDARY OUTCOMES:
Cardiac Magnetic Resonance Imaging | At 30th day after randomization
  Cardiovascular MRI will be performed at 30th day, to detect microvascular obstruction (MO) and intramyocardial hemorrhage (IMH). Infarct size and myocardial strain will also be measured by the method previously described.
Echocardiography | At 30th day after randomization
  echocardiography will be performed within 24h post PCI and at 30th day to assess changes in left ventricular size and function
Myocardial-specific isoenzyme of creatine kinase (CK-MB) enzyme levels peri-PCI | Within 0 to 48 hours after enrollment
  Infarct size is measured by the myocardial-specific isoenzyme of creatine kinase (CK-MB) area under the curve, calculated by the linear-trapezoidal method. If the baseline or last value is missing, the corresponding value will be set to zero. For missing values of intermediate time points, linear interpolation is used.

OTHER OUTCOMES:
Bleeding events: Incidence of bleeding events | Within 0 to 30 dys after randomization
  Incidence of bleeding events, classified by TIMI criteria and GUSTO severity criteria.
Other adverse events | Within 0 to 30 days after randomization
  Including any other adverse events (AEs) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ben He, MD,PhD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Chinese Society of Cardiology of Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. [Guideline of non-ST segment elevation acute coronary syndrome]. Zhonghua Xin Xue Guan Bing Za Zhi. 2012 May;40(5):353-67. No abstract available. Chinese. PMID 22883082
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Roe MT, Ohman EM, Maas AC, Christenson RH, Mahaffey KW, Granger CB, Harrington RA, Califf RM, Krucoff MW. Shifting the open-artery hypothesis downstream: the quest for optimal reperfusion. J Am Coll Cardiol. 2001 Jan;37(1):9-18. doi: 10.1016/s0735-1097(00)01101-3. PMID 11153779
- [Background] Pu J, Shan P, Ding S, Qiao Z, Jiang L, Song W, Du Y, Shen J, Shen L, Jin S, He B. Gender differences in epicardial and tissue-level reperfusion in patients undergoing primary angioplasty for acute myocardial infarction. Atherosclerosis. 2011 Mar;215(1):203-8. doi: 10.1016/j.atherosclerosis.2010.11.019. Epub 2010 Nov 26. PMID 21176835
- [Background] Pu J, Ding S, Shan P, Qiao Z, Song W, Du Y, Shen J, Jin S, He B. Comparison of epicardial and myocardial perfusions after primary coronary angioplasty for ST-elevation myocardial infarction in patients under and over 75 years of age. Aging Clin Exp Res. 2010 Aug;22(4):295-302. doi: 10.1007/BF03337726. Epub 2009 Dec 1. PMID 20009495
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Shen LH, Wan F, Shen L, Ding S, Gong XR, Qiao ZQ, Du YP, Song W, Shen JY, Jin SX, Pu J, Yao TB, Jiang LS, Li WZ, Zhou GW, Liu SW, Han YL, He B. Pharmacoinvasive therapy for ST elevation myocardial infarction in China: a pilot study. J Thromb Thrombolysis. 2012 Jan;33(1):101-8. doi: 10.1007/s11239-011-0657-7. PMID 22094974